CLINICAL TRIAL: NCT02780648
Title: Pilot Study of Respiratory-gated Stereotactic Body Radiation Therapy for Borderline Resectable, Unresectable, or Recurrent/Residual Adenocarcinoma of the Pancreas or Periampullary Region
Brief Title: Respiratory-gated Stereotactic Body Radiation Therapy for Adenocarcinoma of the Pancreas or Periampullary Region
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Robert Miller, Clinical Professor of Radiation Oncology, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUSCC-0565; 1601638414 (Other: Indiana University IRB)
Record Dates: First submitted 2016-05-17; First posted 2016-05-23 (Estimated); Results first posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Pancreatic Neoplasms
Keywords: stereotactic radiotherapy; pancreatic adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Stereotactic Body Radiation (Experimental): Patients will receive 5 fractions of 5 Gy or 6.6 Gy (dose depending upon whether or not they have received prior radiation therapy to the pancreatic region) delivered over a five-day period.
  Interventions: Radiation: Stereotactic Body Radiation

INTERVENTIONS:
Radiation: Stereotactic Body Radiation

SUMMARY:
This is a single center, single arm unblinded prospective study of the safety of pancreatic stereotactic body radiation therapy (SBRT) in patients with unresectable, borderline resectable, or recurrent pancreatic/periampullary cancers who have previously undergone treatment with chemotherapy, surgery, photodynamic therapy, conventionally fractionated radiation treatment, or any combination of these therapies.

Primary Objective

• To estimate rates of acute (within 3 months of treatment) grade 3 or greater gastrointestinal and hematologic toxicity in patients treated with Linac-based SBRT for pancreatic or periampullary cancers who have previously received other treatment.

Secondary Objectives

* To estimate rates of late (> 3 months after treatment) grade 2 gastritis, enteritis, fistula, and ulcer, or any other grade 3 or greater gastrointestinal toxicity in patients treated with Linac-based SBRT for pancreatic or periampullary cancers
* To estimate rates of local progression, overall survival, metastasis-free survival, and progression-free survival in patients with pancreatic or periampullary cancers treated with fractionated Linac-based SBRT.
* To evaluate the ability of Linac-based SBRT to provide pain control in patients with pain related to a pancreatic or periampullary tumor.
* To evaluate quality of life in patients undergoing treatment with Linac-based SBRT for pancreatic or periampullary cancers.

DETAILED DESCRIPTION:
Patients will receive 5 fractions of 5 gray (Gy) or 6.6 Gy delivered over a five-day period based on whether or not they have received prior radiation therapy to the pancreatic region. Treatment may be delivered over 2 weeks, provided that the patient receives at least 2 fractions per week. Initial patient positioning will be based on volumetric kV (cone-beam computerized tomography) imaging with shifts to bony anatomy as appropriate. Orthogonal kV/MV or kV/kV projection imaging will be used to verify the location of the fiducials prior to delivery of the first treatment beam. A secondary shift based on the location of fiducials may be utilized, as indicated by the position of the fiducials. For free-breathing treatments, kV fluoroscopic images should be obtained to confirm the anticipated position of these fiducials during the entire respiratory cycle. Active monitoring of treatment delivery accuracy will be accomplished using kV and/or MV projection imaging, either immediately before or during all (or a subset of) treatment fields. Patient-specific dosimetric quality assurance (QA) will be performed as per standard practice in the Department of Radiation Oncology, Indiana University School of Medicine.

ELIGIBILITY:
Inclusion Criteria

* Age >18 years.
* Karnofsky Performance Status >70%
* Histologically confirmed adenocarcinoma of the pancreas or ampulla of Vater; at least the majority of the histopathologic specimen must be identified as adenocarcinoma as opposed to another histologic subtype. In patients with a diagnosis of recurrent disease (based on radiographic progression and/or rising CA19-9 levels) and a history of a biopsy-proven adenocarcinoma of the pancreas or the ampulla of Vater, repeat biopsy of the recurrence site is not required for participation of the trial.
* Pancreatic or periampullary tumors must be less than 8.0 cm in greatest axial dimension at the time of treatment planning.
* Patients who have been treated with any combination of surgical resection and neoadjuvant/adjuvant conventional chemoradiation therapy for resectable disease or conventional chemoradiation as definitive treatment for unresectable or borderline resectable disease are eligible for the study, provided that at least 180 days have elapsed since completing any previous radiation treatment. Patients who have been receiving continued chemotherapy following their initial radiation treatment are eligible regardless of when the most recent chemotherapy was received. Those patients who have received prior radiation therapy will constitute Cohort A and will receive stereotactic body radiation (SBRT) as 5 gray (Gy) x 5.
* Patients who have not previously undergone radiation therapy can have a history of treatment with either chemotherapy (for unresectable/borderline resectable disease) or any combination of surgery and chemotherapy (for resectable disease). Patients with no history of prior radiation treatment will constitute Cohort B and will receive SBRT as 6.6 Gy x 5. Please note that patients must have received at least two cycles of chemotherapy (with selection of drugs at the discretion of the treating oncologist) before SBRT treatment on protocol.
* Acceptable organ and marrow function as defined below (within 2 weeks prior to radiotherapy):

  * Leukocytes >3,000/μL
  * Absolute neutrophil count >1,500μL
  * Platelets >100,000/μL
  * Total Bilirubin ≤1.5x institutional upper limit of normal
  * Aspartate transaminase (AST(SGOT))/Alanine transaminase (ALT(SGPT)) <2.5x institutional upper limit of normal
  * Creatinine ≤ institutional upper limit of normal OR creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Ability to understand and the willingness to sign a written informed consent document.
* Life expectancy > 3 months.
* Radio-opaque markers must be present within the tumor bed. In patients who have undergone surgical resection, radio-opaque surgical clips within the tumor bed can be used as fiducials. Patients without surgical clips in the tumor bed must be able to have fiducials placed endoscopically, laparoscopically, or through a CT- or ultrasound-guided technique. If not, the tumor must be posterior and adjacent to the aorta, and treatment will only be permitted at the discretion of the Principal Investigator.

Exclusion Criteria

* Age < 18 years.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (or infections requiring systemic antibiotic treatment), active upper GI ulceration or hemorrhage, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Any concurrent malignancy other than non-melanoma skin cancer, non-invasive bladder cancer, early stage prostate cancer, or carcinoma in situ of the cervix. Patients with a previous non-pancreatic, non-periampullary malignancy without evidence of disease for > 5 years will be allowed to enter the trial.
* Pregnant and breastfeeding women are excluded as are women of child-bearing potential who are unwilling or unable to use an acceptable method of birth control (hormonal or barrier method of birth control; abstinence) to avoid pregnancy for the duration of the study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Women who are not post-menopausal (as defined in Appendix III) and have a positive urine or serum pregnancy test or refuse to take a pregnancy test.
* Patients with a life expectancy of < 3 months.
* Patients with metastatic disease.
* Patients with evidence of gross tumor invasion into the lumen of the stomach or small bowel are not eligible; if imaging suggests luminal invasion of tumor, this must be ruled out endoscopically before the patient can be enrolled on study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2025-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Miller, MD, Principal Investigator — Indiana University School of Medicine, Indiana University Simon Cancer Center
Locations (2):
- United States (2):
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Patients who have received prior radiation therapy and received Stereotactic Body Radiation Therapy (SBRT) as 5 Gy x 5.
- Cohort B: Patients with no history of prior radiation treatment and who received SBRT as 6.6 Gy x 5
Period: Overall Study
Arm/Group | Cohort A | Cohort B
Started | 3 | 33
Completed | 2 | 33
Not Completed | 1 | 0
Not completed — Disease Progression | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 3 | 33 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (7.2) | 66.5 (9.6) | 66.3 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 18 | 20
  Male | 1 | 15 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 31 | 33
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 3 | 27 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 33 | 36

OUTCOME MEASURES:

1. Primary Outcome: Acute Toxicity Rates of Grade 3 or Greater Gastrointestinal and Hematologic Toxicities (as Raw Percentage)
Description: Measures include the percentage of patients who experienced the toxicity with a grade of 3 or higher. Only those adverse events that were related to stereotactic body radiation therapy (SBRT) were considered. Patients were considered at risk for an adverse event if they started SBRT treatment. Toxicities per Common Terminology Criteria for Adverse Events (CTCAE) 4.0.
Time Frame: Up to 90 days after treatment
Population: Includes all patients in cohorts A and B who met eligibility criteria for primary outcome measure.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- All Eligible Participants: The two cohorts were combined since the safety profile was expected to be similar.
  Cohort A included patients who have received prior radiation therapy and received Stereotactic Body Radiation Therapy (SBRT) as 5 Gy x 5. Cohort B included patients with no history of prior radiation treatment and who received SBRT as 6.6 Gy x 5.
Arm/Group | All Eligible Participants
Number analyzed (Participants) | 36
percentage of participants
  Hematologic: Lymphocyte Count Decreased | 13.89 [4.41 to 23.37]
  Hematologic: White Blood Cell Decreased | 0.00 [0.00 to 0.00]
  Gastrointestinal: Nausea | 2.78 [0.00 to 7.28]
  Gastrointestinal: Abdominal Pain | 0.00 [0.00 to 0.00]
  Gastrointestinal: Diarrhea | 0.00 [0.00 to 0.00]
  Gastrointestinal: Bloating | 0.00 [0.00 to 0.00]
  Gastrointestinal: Flatulence | 0.00 [0.00 to 0.00]
  Gastrointestinal: Gastritis | 0.00 [0.00 to 0.00]
  Gastrointestinal: Vomiting | 2.78 [0.00 to 7.28]

2. Secondary Outcome: Late, Treatment-related Toxicity Rates of Gastritis, Enteritis, Fistula, and Ulcer, or Any Other Gastrointestinal Toxicity (as Raw Percentage)
Description: Measures include the percentage of patients who experienced the toxicity with a grade of 2 or higher. Only those adverse events that were related to stereotactic body radiation therapy (SBRT) were considered. Patients were considered at risk for an adverse event if they started SBRT treatment. Toxicities per Common Terminology Criteria for Adverse Events (CTCAE) 4.0.
Time Frame: 90 or more days after treatment, up to 7 years
Population: Includes those patients who were determined to be eligible for the secondary outcome measures.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | All Eligible Participants
Number analyzed (Participants) | 36
percentage of participants
  Gastritis | 0.00 [0.00 to 0.00]
  Enteritis | 0.00 [0.00 to 0.00]
  Fistula | 0.00 [0.00 to 0.00]
  Ulcer | 0.00 [0.00 to 0.00]
  Diarrhea | 0.00 [0.00 to 0.00]
  Vomiting | 0.00 [0.00 to 0.00]

3. Secondary Outcome: Overall Survival
Description: This measure reports the overall survival probability from the Kaplan Meier method. The survival time was calculated from the date of treatment start to the date of death and patients who did not expire were censored at their last date known alive.
Time Frame: 1 year after treatment
Population: Includes patients in Cohort B who were considered eligible for the outcome analyses.
Measure: Number (90% Confidence Interval); unit: survival probability
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 0 | 33
survival probability |  | .4849 [.3368 to .6178]

4. Secondary Outcome: Progression-Free Survival
Description: This measure represents the progression-free survival at one-year following treatment start. The survival time was calculated from the date of treatment start to the date of progression or death. Patients who did not experience progression were censored at their last known date alive.
Time Frame: 1 year after treatment
Population: Includes patients in cohort B who were determined to be eligible for the secondary objectives.
Measure: Number (90% Confidence Interval); unit: survival probability
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 0 | 33
survival probability |  | .3939 [.2557 to .5293]

5. Secondary Outcome: Metastasis-Free Survival
Description: This represents the metastasis-free survival at one-year following treatment start. The survival time was calculated from the date of treatment start to the date of metastasis or death. Patients who did not experience metastasis or death were censored at their last known date alive.
Time Frame: 1 year after treatment
Population: Includes patients in Cohort B who were determined to be eligible for the secondary outcomes analyses.
Measure: Number (90% Confidence Interval); unit: survival probability
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 0 | 33
survival probability |  | .4846 [.3368 to .6178]

6. Secondary Outcome: Wong-Baker FACES Pain Rating Score
Description: Measured with the Wong-Baker FACES 0-10 scale where higher scores indicate more pain. Patients self-reported the score before (baseline), during (weeks 1 and 2), and after (1 and 3 months) treatment. Scores collected during treatment (weeks 1 and 2) were averaged to create a composite "during treatment" score. Similarly, scores collected after treatment (months 1 and 3) were averaged to create a composite "after treatment" score.
Time Frame: Baseline (before treatment), Week 1 (during treatment), Week 2 (during treatment), Month 1 (after treatment), and Month 3 (after treatment)
Population: Includes all patients who were determined to be eligible for the secondary outcomes.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 3 | 33
score on a scale
  Before Treatment Score | 1.00 [0.00 to 2.50] | 2.00 [0.00 to 4.00]
  During Treatment Score | 2.00 [1.00 to 2.00] | 0.00 [0.00 to 2.00]
  After Treatment Score | 2.00 [0.00 to 2.00] | 0.00 [0.00 to 4.00]
Statistical Analysis 1: Comparison: Cohort B; For Cohort B, pain scores were compared across treatment phase (before, during, and after) using ordinal logistic regression models with repeated measures; Test type: Other; p = 0.824, Mixed Models Analysis — This p-value represents the type III p-value for overall treatment phase variable significance. An a priori alpha level of 0.05 was used to determine statistical significance

7. Secondary Outcome: Quality of Life Scores - Global Health Status / Quality of Life
Description: Patients completed the EORTC Quality of Life (QOL)-Q (QLQ-C30 Version 3) questionnaire before treatment, during treatment, and after treatment. The questionnaire includes 30 questions to assess the quality of life in cancer patients. The Global Health Status / Quality of Life composite score was calculated by combining the scores for questions 29 and 30 and calculating Score = {(RS -1) range}×100. Responses for questions 29 and 30 ranged from 1 to 7 with 1 indicating "Very Poor" and 7 indicating "Excellent". Higher scores indicate a better quality of life with a minimum composite score of 0 and a maximum composite score of 100. Scores collected during treatment (weeks 1 and 2) were averaged to create a composite "during treatment" score. Similarly, scores collected after treatment (months 1, 3, 6, 9, and 12) were averaged to create a composite "after treatment" score.
Time Frame: Baseline (before treatment), 1 week (during treatment), 2 weeks (during treatment), 1 month (after treatment), 3 months (after treatment), 6 months (after treatment), 9 months (after treatment), and 12 months (after treatment)
Population: Includes patients who were eligible for the secondary outcomes.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 3 | 33
score on a scale
  Global Health Status - Before Treatment: number analyzed (Participants) | 2 | 25
  Global Health Status - Before Treatment | 83.33 [83.33 to 83.33] | 75.00 [50.00 to 83.33]
  Global Health Status - During Treatment: number analyzed (Participants) | 2 | 30
  Global Health Status - During Treatment | 83.33 [83.33 to 83.33] | 66.67 [50.00 to 83.33]
  Global Health Status - After Treatment: number analyzed (Participants) | 2 | 28
  Global Health Status - After Treatment | 79.17 [43.75 to 83.33] | 70.83 [50.00 to 83.33]
Statistical Analysis 1: Comparison: Cohort B; The null hypothesis was that there was no difference in composite global health status / quality of life scores across treatment phase; Test type: Other — Ordinal logistic regression models with repeated measures to account for multiple patient surveys were fit with treatment phase (before treatment, during treatment, and after treatment) as the predictor and composite global health status / quality of life score as the outcome; p = 0.270, Regression, Logistic — The a priori threshold for statistical significance was 0.05. P-value represents the omnibus p-value for treatment phase in the repeated-measures ordinal logistic regression model

8. Secondary Outcome: Quality of Life Scores - Functional Scales
Description: Patients completed the EORTC Quality of Life (QOL)-Q (QLQ-C30 Version 3) questionnaire before treatment, during treatment, and after treatment. The questionnaire includes 30 questions to assess the quality of life in cancer patients. The Functional scales composite scores were calculated by combining the scores for the relevant questions and calculating Score = {1 - ((RS -1) / range)}×100. The response options for each question were "1-Not at all", "2-A little", "3-Quite a bit", and "4-Very Much". Higher scores indicate a high/healthy level of functioning with a minimum composite score of 0 and a maximum composite score of 100. In each category, scores collected during treatment (weeks 1 and 2) were averaged to create a composite "during treatment" score. Similarly, scores collected after treatment (months 1, 3, 6, 9, and 12) were averaged to create a composite "after treatment" score.
Time Frame: as for outcome 7
Population: Includes patients who were eligible for the secondary outcomes.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 3 | 33
score on a scale
  Physical Functioning - Before Treatment: number analyzed (Participants) | 2 | 25
  Physical Functioning - Before Treatment | 76.67 [71.67 to 81.67] | 93.33 [86.67 to 100.00]
  Physical Functioning - During Treatment: number analyzed (Participants) | 2 | 30
  Physical Functioning - During Treatment | 86.67 [86.67 to 88.33] | 86.67 [73.33 to 93.33]
  Physical Functioning - After Treatment: number analyzed (Participants) | 2 | 28
  Physical Functioning - After Treatment | 80.00 [73.33 to 96.67] | 86.67 [80.00 to 100.00]
  Role Functioning - Before Treatment: number analyzed (Participants) | 2 | 25
  Role Functioning - Before Treatment | 50.00 [41.67 to 58.33] | 83.33 [66.67 to 100.00]
  Role Functioning - During Treatment: number analyzed (Participants) | 2 | 30
  Role Functioning - During Treatment | 75.00 [66.67 to 83.33] | 83.33 [66.67 to 100.00]
  Role Functioning - After Treatment: number analyzed (Participants) | 2 | 28
  Role Functioning - After Treatment | 75.00 [41.67 to 95.83] | 100.00 [66.67 to 100.00]
  Emotional Functioning - Before Treatment: number analyzed (Participants) | 2 | 25
  Emotional Functioning - Before Treatment | 75.00 [70.83 to 79.17] | 83.33 [66.67 to 91.67]
  Emotional Functioning - During Treatment: number analyzed (Participants) | 2 | 30
  Emotional Functioning - During Treatment | 83.33 [81.25 to 83.33] | 91.67 [75.00 to 100.00]
  Emotional Functioning - After Treatment: number analyzed (Participants) | 2 | 28
  Emotional Functioning - After Treatment | 75.00 [68.75 to 81.25] | 83.33 [72.92 to 100.00]
  Cognitive Functioning - Before Treatment: number analyzed (Participants) | 2 | 25
  Cognitive Functioning - Before Treatment | 91.67 [87.50 to 95.83] | 83.33 [66.67 to 100.00]
  Cognitive Functioning - During Treatment: number analyzed (Participants) | 2 | 30
  Cognitive Functioning - During Treatment | 100.00 [100.00 to 100.00] | 83.33 [83.33 to 100.00]
  Cognitive Functioning - After Treatment: number analyzed (Participants) | 2 | 28
  Cognitive Functioning - After Treatment | 83.33 [70.83 to 95.83] | 83.33 [79.17 to 100.00]
  Social Functioning - Before Treatment: number analyzed (Participants) | 2 | 25
  Social Functioning - Before Treatment | 33.33 [33.33 to 33.33] | 66.67 [50.00 to 83.33]
  Social Functioning - During Treatment: number analyzed (Participants) | 2 | 30
  Social Functioning - During Treatment | 83.33 [62.50 to 100.00] | 66.67 [50.00 to 100.00]
  Social Functioning - After Treatment: number analyzed (Participants) | 2 | 28
  Social Functioning - After Treatment | 66.67 [54.17 to 91.67] | 83.33 [66.67 to 100.00]
Statistical Analysis 1: Comparison: Cohort B; The null hypothesis was that there was no difference in composite physical functioning composite scores across treatment phase; Test type: Other — Ordinal logistic regression models with repeated measures to account for multiple patient surveys were fit with treatment phase (before treatment, during treatment, and after treatment) as the predictor and composite physicial functioning composite score as the outcome; p = 0.179, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Cohort B; The null hypothesis was that there was no difference in composite role functioning composite scores across treatment phase; Test type: Other — Ordinal logistic regression models with repeated measures to account for multiple patient surveys were fit with treatment phase (before treatment, during treatment, and after treatment) as the predictor and composite role functioning composite score as the outcome; p = 0.789, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: Cohort B; The null hypothesis was that there was no difference in composite emotional functioning composite scores across treatment phase; Test type: Other — Ordinal logistic regression models with repeated measures to account for multiple patient surveys were fit with treatment phase (before treatment, during treatment, and after treatment) as the predictor and composite emotional functioning composite score as the outcome; p = 0.303, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: Cohort B; The null hypothesis was that there was no difference in composite cognitive functioning composite scores across treatment phase; Test type: Other — Ordinal logistic regression models with repeated measures to account for multiple patient surveys were fit with treatment phase (before treatment, during treatment, and after treatment) as the predictor and composite cognitive functioning composite score as the outcome; p = 0.989, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 5: Comparison: Cohort B; The null hypothesis was that there was no difference in composite social functioning composite scores across treatment phase; Test type: Other — Ordinal logistic regression models with repeated measures to account for multiple patient surveys were fit with treatment phase (before treatment, during treatment, and after treatment) as the predictor and composite social functioning composite score as the outcome; p = 0.436, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]

9. Secondary Outcome: Quality of Life Scores - Symptom Scales
Description: Patients completed the EORTC Quality of Life (QOL)-Q (QLQ-C30 Version 3) questionnaire before treatment, during treatment, and after treatment. The questionnaire includes 30 questions to assess the quality of life in cancer patients. The Symptom scales composite scores were calculated by combining the scores for the relevant questions and calculating Score = {(RS -1) range}×100. The response options for each question were "1-Not at all", "2-A little", "3-Quite a bit", and "4-Very Much". Higher scores indicate a high level of symptomatology / problems with a minimum composite score of 0 and a maximum composite score of 100. In each category, scores collected during treatment (weeks 1 and 2) were averaged to create a composite "during treatment" score. Similarly, scores collected after treatment (months 1, 3, 6, 9, and 12) were averaged to create a composite "after treatment" score.
Time Frame: as for outcome 7
Population: Includes patients who were eligible for the secondary outcomes.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 3 | 33
score on a scale
  Fatigue - Before Treatment: number analyzed (Participants) | 2 | 25
  Fatigue - Before Treatment | 44.44 [33.33 to 55.56] | 33.33 [25.00 to 44.44]
  Fatigue - During Treatment: number analyzed (Participants) | 2 | 30
  Fatigue - During Treatment | 33.33 [33.33 to 33.33] | 33.33 [22.22 to 55.56]
  Fatigue - After Treatment: number analyzed (Participants) | 2 | 28
  Fatigue - After Treatment | 44.44 [33.33 to 72.22] | 33.33 [11.11 to 44.44]
  Nausea and Vomiting - Before Treatment: number analyzed (Participants) | 2 | 25
  Nausea and Vomiting - Before Treatment | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 16.67]
  Nausea and Vomiting - During Treatment: number analyzed (Participants) | 2 | 30
  Nausea and Vomiting - During Treatment | 8.33 [0.00 to 16.67] | 16.67 [0.00 to 16.67]
  Nausea and Vomiting - After Treatment: number analyzed (Participants) | 2 | 28
  Nausea and Vomiting - After Treatment | 25.00 [16.67 to 33.33] | 0.00 [0.00 to 16.67]
  Pain - Before Treatment: number analyzed (Participants) | 2 | 25
  Pain - Before Treatment | 41.67 [37.50 to 45.83] | 16.67 [0.00 to 33.33]
  Pain - During Treatment: number analyzed (Participants) | 2 | 30
  Pain - During Treatment | 16.67 [16.67 to 20.83] | 33.33 [0.00 to 50.00]
  Pain - After Treatment: number analyzed (Participants) | 2 | 28
  Pain - After Treatment | 33.33 [20.83 to 58.33] | 16.67 [0.00 to 50.00]
  Dyspnea - Before Treatment: number analyzed (Participants) | 2 | 25
  Dyspnea - Before Treatment | 16.67 [8.33 to 25.00] | 0.00 [0.00 to 0.00]
  Dyspnea - During Treatment: number analyzed (Participants) | 2 | 30
  Dyspnea - During Treatment | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Dyspnea - After Treatment: number analyzed (Participants) | 2 | 28
  Dyspnea - After Treatment | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 33.33]
  Insomnia - Before Treatment: number analyzed (Participants) | 2 | 25
  Insomnia - Before Treatment | 33.33 [16.67 to 50.00] | 33.33 [0.00 to 33.33]
  Insomnia - During Treatment: number analyzed (Participants) | 2 | 30
  Insomnia - During Treatment | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 33.33]
  Insomnia - After Treatment: number analyzed (Participants) | 2 | 28
  Insomnia - After Treatment | 16.67 [0.00 to 33.33] | 0.00 [0.00 to 33.33]
  Appetite Loss - Before Treatment: number analyzed (Participants) | 2 | 25
  Appetite Loss - Before Treatment | 16.67 [8.33 to 25.00] | 0.00 [0.00 to 33.33]
  Appetite Loss - During Treatment: number analyzed (Participants) | 2 | 30
  Appetite Loss - During Treatment | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 33.33]
  Appetite Loss - After Treatment: number analyzed (Participants) | 2 | 28
  Appetite Loss - After Treatment | 16.67 [0.00 to 58.33] | 0.00 [0.00 to 33.33]
  Constipation - Before Treatment: number analyzed (Participants) | 2 | 25
  Constipation - Before Treatment | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 33.33]
  Constipation - During Treatment: number analyzed (Participants) | 2 | 30
  Constipation - During Treatment | 0.00 [0.00 to 8.33] | 16.67 [0.00 to 33.33]
  Constipation - After Treatment: number analyzed (Participants) | 2 | 28
  Constipation - After Treatment | 0.00 [0.00 to 25.00] | 0.00 [0.00 to 0.00]
  Diarrhea - Before Treatment: number analyzed (Participants) | 2 | 25
  Diarrhea - Before Treatment | 0.00 [0.00 to 0.00] | 16.67 [0.00 to 33.33]
  Diarrhea - During Treatment: number analyzed (Participants) | 2 | 30
  Diarrhea - During Treatment | 16.67 [0.00 to 33.33] | 0.00 [0.00 to 33.33]
  Diarrhea - After Treatment: number analyzed (Participants) | 2 | 28
  Diarrhea - After Treatment | 16.67 [0.00 to 33.33] | 33.33 [0.00 to 33.33]
  Financial Difficulties - Before Treatment: number analyzed (Participants) | 2 | 25
  Financial Difficulties - Before Treatment | 66.67 [66.67 to 66.67] | 33.33 [0.00 to 66.67]
  Financial Difficulties - During Treatment: number analyzed (Participants) | 2 | 30
  Financial Difficulties - During Treatment | 16.67 [0.00 to 33.33] | 33.33 [0.00 to 66.67]
  Financial Difficulties - After Treatment: number analyzed (Participants) | 2 | 28
  Financial Difficulties - After Treatment | 33.33 [8.33 to 58.33] | 33.33 [0.00 to 33.33]
Statistical Analysis 1: Comparison: Cohort B; The null hypothesis was that there was no difference in composite fatigue symptom scores across treatment phase; Test type: Other — Ordinal logistic regression models with repeated measures to account for multiple patient surveys were fit with treatment phase (before treatment, during treatment, and after treatment) as the predictor and composite fatigue symptom score as the outcome; p = 0.659, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Cohort B; The null hypothesis was that there was no difference in composite nausea and vomiting symptom scores across treatment phase; Test type: Other — Ordinal logistic regression models with repeated measures to account for multiple patient surveys were fit with treatment phase (before treatment, during treatment, and after treatment) as the predictor and composite nausea and vomiting symptom score as the outcome; p = 0.295, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: Cohort B; The null hypothesis was that there was no difference in composite pain symptom scores across treatment phase; Test type: Other — Ordinal logistic regression models with repeated measures to account for multiple patient surveys were fit with treatment phase (before treatment, during treatment, and after treatment) as the predictor and composite pain symptom score as the outcome; p = 0.299, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: Cohort B; The null hypothesis was that there was no difference in composite dyspnea symptom scores across treatment phase; Test type: Other — Ordinal logistic regression models with repeated measures to account for multiple patient surveys were fit with treatment phase (before treatment, during treatment, and after treatment) as the predictor and composite dyspnea symptom score as the outcome; p = 0.794, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 5: Comparison: Cohort B; The null hypothesis was that there was no difference in composite insomnia symptom scores across treatment phase; Test type: Other — Ordinal logistic regression models with repeated measures to account for multiple patient surveys were fit with treatment phase (before treatment, during treatment, and after treatment) as the predictor and composite insomnia symptom score as the outcome; p = 0.450, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 6: Comparison: Cohort B; The null hypothesis was that there was no difference in composite appetite loss symptom scores across treatment phase; Test type: Other — Ordinal logistic regression models with repeated measures to account for multiple patient surveys were fit with treatment phase (before treatment, during treatment, and after treatment) as the predictor and composite appetite loss symptom score as the outcome; p = 0.389, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 7: Comparison: Cohort B; The null hypothesis was that there was no difference in composite constipation symptom scores across treatment phase; Test type: Other — Ordinal logistic regression models with repeated measures to account for multiple patient surveys were fit with treatment phase (before treatment, during treatment, and after treatment) as the predictor and composite constipation symptom score as the outcome; p = 0.011, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]; The odds of having a higher constipation symptom composite score after treatment were less than during or before treatment
Statistical Analysis 8: Comparison: Cohort B; The null hypothesis was that there was no difference in composite diarrhea symptom scores across treatment phase; Test type: Other — Ordinal logistic regression models with repeated measures to account for multiple patient surveys were fit with treatment phase (before treatment, during treatment, and after treatment) as the predictor and composite diarrhea symptom score as the outcome; p = 0.101, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 9: Comparison: Cohort B; The null hypothesis was that there was no difference in composite financial difficulty symptom scores across treatment phase; Test type: Other — Ordinal logistic regression models with repeated measures to account for multiple patient surveys were fit with treatment phase (before treatment, during treatment, and after treatment) as the predictor and composite financial difficulty symptom score as the outcome; p = 0.306, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]

ADVERSE EVENTS:
Time Frame: 7 years from start of treatment
Arm/Group | Cohort A | Cohort B
All-Cause Mortality (participants affected / at risk) | 3/3 | 33/33
Serious Adverse Events (participants affected / at risk) | 3/3 | 33/33
Other Adverse Events (participants affected / at risk) | 3/3 | 24/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=3) | Cohort B (N=33)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Hepatobiliary disorders - Other, sp (Hepatobiliary disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Abdominal infection (Infections and infestations) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 2
Allergic reaction (Immune system disorders) | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 4
Biliary tract infection (Infections and infestations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 1
Duodenal infection (Infections and infestations) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Esophageal infection (Infections and infestations) | 0 | 1
Fever (General disorders and administration site conditions) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Hematoma (Vascular disorders) | 0 | 1
Hypothermia (General disorders and administration site conditions) | 0 | 1
INR increased (Investigations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Pain (General disorders and administration site conditions) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=3) | Cohort B (N=33)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 4 (4)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 20 (39)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 13 (22)
Alkaline phosphatase increased (Investigations) | 1 (1) | 8 (11)
Allergic reaction (Immune system disorders) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 12 (24)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 4 (10)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 15 (24)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 8 (8)
Biliary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (2) | 5 (5)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 2 (4)
Blood bilirubin increased (Investigations) | 0 (0) | 10 (20)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
CPK increased (Investigations) | 0 (0) | 1 (1)
Chills (General disorders and administration site conditions) | 1 (1) | 3 (3)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (5)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 10 (13)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders and administration site conditions) | 0 (0) | 5 (5)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Esophageal infection (Infections and infestations) | 0 (0) | 1 (1)
Fatigue (General disorders and administration site conditions) | 2 (2) | 17 (22)
Fever (General disorders and administration site conditions) | 1 (1) | 6 (6)
Flatulence (Gastrointestinal disorders) | 1 (2) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Gait disturbance (General disorders and administration site conditions) | 0 (0) | 2 (2)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 3 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Hallucinations (Psychiatric disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 2 (3)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 2 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 5 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 5 (7)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypothermia (General disorders and administration site conditions) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 2 (3)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1) | 2 (5)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Localized edema (General disorders and administration site conditions) | 0 (0) | 2 (2)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (4) | 16 (26)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (3) | 12 (17)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 3 (5)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain (General disorders and administration site conditions) | 0 (0) | 3 (6)
Pancreatic enzymes decreased (Investigations) | 0 (0) | 2 (3)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 6 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)
Urine output decreased (Investigations) | 0 (0) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (7)
Weight gain (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 6 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT02780648/Prot_SAP_000.pdf